CLINICAL TRIAL: NCT02621580
Title: A 24-Month Cohort Study Assessing the Nature and the Time Course of Structural and Functional Changes to the Retina Following PASCAL Photocoagulation in Proliferative Diabetic Retinopathy Patients
Brief Title: Investigating the Structural and Functional Changes to the Retina Following PRP in Diabetic Retinopathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103197
Record Dates: First submitted 2015-11-27; First posted 2015-12-03 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Retinopathy
Keywords: Panretinal Photocoagulation
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients with type 1 or type 2 diabetes mellitus (according to ADA or WHO guidelines) that have severe preproliferative or proliferative diabetic retinopathy and do not require laser or anti-VEGF treatment in at least one eye.
- Treatment: Pan-Retinal Photocoagulation (Experimental): Patients with type 1 or type 2 diabetes mellitus (according to ADA or WHO guidelines) that have severe preproliferative or proliferative diabetic retinopathy and require PRP laser in at least one eye.
  Interventions: Device: Pan-Retinal Photocoagulation

INTERVENTIONS:
Device: Pan-Retinal Photocoagulation — Diabetic retinopathy does not usually impair sight until the development of long-term complications, including proliferative retinopathy, a condition in which abnormal new blood vessels may rupture and bleed inside the eye. When this advanced stage of retinopathy occurs, pan-retinal photocoagulation is usually recommended.
  During this procedure, a special laser is used to make tiny burns that seal the retina and stop vessels from growing and leaking. Hundreds of tiny spots of laser are placed in the retina to reduce the risk of vitreous haemorrhage and retinal detachment.
  Arms: Treatment: Pan-Retinal Photocoagulation

SUMMARY:
Laser therapy is an established method to stabilize and control proliferative diabetic eye disease. Questions on the long-term effect on the retina from these treatments remain to be answered. The purpose of the study was to evaluate changes in the retina following panretinal photocoagulation (PRP) over time, using structural and functional diagnostic tests.

DETAILED DESCRIPTION:
Diabetic retinopathy is the most common cause of adult-acquired retinal vascular disease. Diabetic retinopathy is estimated to affect more than 100 million adults, and is the leading cause of blindness worldwide.

Over the past 30 years, epidemiological studies and clinical trials have shown that early detection through annual eye exams, intensive glucose and blood pressure control, and timely laser photocoagulation could prevent visual loss. More recently, a variety of newer ocular treatments and medications have been introduced, such as the use of the PASCAL photocoagulation laser system, and various anti-vascular endothelial growth factor therapies. While these treatments have revolutionized how diabetic retinopathy patients are managed clinically, questions on appropriate patient selection and the long-term efficacy and safety of these treatments remain to be answered.

The purpose of this study is to focus on studying the nature and the time course over 2 years of structural and functional changes to the retina following PASCAL photocoagulation in severe preproliferative or proliferative diabetic retinopathy patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient's greater than 18 years of age who have signed an informed consent.
* Patients with type 1 or type 2 diabetes mellitus (according to ADA or WHO guidelines) that have severe preproliferative or proliferative diabetic retinopathy and require PRP surgery in at least one eye.
* Adequate pupil dilation and clear media to perform laser photocoagulation, HRT, OCT and visual field testing.

Exclusion Criteria:

* Advanced lens opacity (Lens opacity that excludes the ability to capture data)
* Prior PRP within the past year
* Focal laser within one year of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
The rate of structural and functional changes to the retinal thickness following PASCAL PRP in severe PDR patients, assessed by optical coherence tomography. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Hutnik, MD, PhD, Principal Investigator — Western University

REFERENCES:
- [Background] Klein R. Prevention of visual loss from diabetic retinopathy. Surv Ophthalmol. 2002 Dec;47 Suppl 2:S246-52. doi: 10.1016/s0039-6257(02)00388-0. PMID 12507626
- [Background] Lim MC, Tanimoto SA, Furlani BA, Lum B, Pinto LM, Eliason D, Prata TS, Brandt JD, Morse LS, Park SS, Melo LA Jr. Effect of diabetic retinopathy and panretinal photocoagulation on retinal nerve fiber layer and optic nerve appearance. Arch Ophthalmol. 2009 Jul;127(7):857-62. doi: 10.1001/archophthalmol.2009.135. PMID 19597104
- [Background] Kim HY, Cho HK. Peripapillary retinal nerve fiber layer thickness change after panretinal photocoagulation in patients with diabetic retinopathy. Korean J Ophthalmol. 2009 Mar;23(1):23-6. doi: 10.3341/kjo.2009.23.1.23. Epub 2009 Mar 9. PMID 19337475
- [Background] Muqit MM, Marcellino GR, Henson DB, Fenerty CH, Stanga PE. Randomized clinical trial to evaluate the effects of Pascal panretinal photocoagulation on macular nerve fiber layer: Manchester Pascal Study report 3. Retina. 2011 Sep;31(8):1699-707. doi: 10.1097/IAE.0b013e318207d188. PMID 21478808